CLINICAL TRIAL: NCT02530099
Title: Simulation-based Training of Operating Assistants: Procedure- Versus Camera Navigation Training - a Randomized Controlled Trial Examining Clinical Transfer
Brief Title: Simulation-based Training of Operating Assistants: Procedure- Versus Camera Navigation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Cecilia Nilsson, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: CN-Trial
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Laparoscopic Simulation Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Receive no training.
- CN-group (Experimental): Receive basic camera navigation training.
  Interventions: Procedure: CN-group
- Procedure-group (Experimental): Receive training on a laparoscopic procedure.
  Interventions: Procedure: Procedure-group

INTERVENTIONS:
Procedure: CN-group — Time limited simulation based training on camera navigation tasks on a virtual reality-simulator.
  Arms: CN-group
Procedure: Procedure-group — Time limited simulation based training on laparoscopic procedure on a virtual reality-simulator.
  Arms: Procedure-group

SUMMARY:
Often the less experienced as medical students are charged with the role as camera navigator and assistant during laparoscopic surgery. Camera navigation is generally considered an easy skill, but it requires specific psychomotor and visuospatial skills. Simulation-based training can improve surgical skills, but little is known on how to optimally structure a training program to acquire camera navigation skills. The objective of this trial is to examine if simulation-based laparoscopic camera navigation skills transfer to the operating room after practicing one of two fundamentally different laparoscopic tasks on a simulator. The first group practice a procedure on a virtual reality simulator, the second group practice camera navigation on a virtual reality simulator and the third group receive no training. All participants are tested as camera navigators and assistants during a procedure in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Medical students on the 4th, 5th or 6th semester, enrolled at The Faculty of Health Science, University of Copenhagen
* Signed informed consent

Exclusion Criteria:

* Previous participation in trials involving simulated laparoscopic training.
* Experience with laparoscopy surgery (having performed minimum one laparoscopic procedure as primary surgeon or as a surgical assistant).
* No informed consent.
* Does not speak Danish on a conversational level.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Surgeons' rating on camera navigation performance during a procedure in the operating room. | up to 1-3 weeks post training

SECONDARY OUTCOMES:
Score on the intrinsic motivation inventory-scale | 2 months
  An expression of motivation as a surgical assistant and camera navigation after completion of the procedure in the OR

REFERENCES:
- [Derived] Nilsson C, Sorensen JL, Konge L, Westen M, Stadeager M, Ottesen B, Bjerrum F. Simulation-based camera navigation training in laparoscopy-a randomized trial. Surg Endosc. 2017 May;31(5):2131-2139. doi: 10.1007/s00464-016-5210-5. Epub 2016 Oct 21. PMID 27770252